CLINICAL TRIAL: NCT05625126
Title: Evaluation of a Rumination Intervention for Individuals With PTSD: A Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford Health NHS Foundation Trust (Other Government); Berkshire Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 318316
Record Dates: First submitted 2022-11-02; First posted 2022-11-22 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Posttraumatic Stress Disorder; Rumination - Thoughts
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Multiple baseline case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rumination Invervention - 3 week baseline (Experimental): Baseline measures will be collected weekly for 3 weeks.
  All participants will then receive a one-session online Rumination Intervention for PTSD with a follow-up call to clarify/solidify learning.
  Interventions: Other: Rumination Intervention for individuals with PTSD
- Rumination Invervention - 5 week baseline (Experimental): Baseline measures will be collected weekly for 5 weeks.
  All participants will then receive a one-session online Rumination Intervention for PTSD with a follow-up call to clarify/solidify learning.
  Interventions: Other: Rumination Intervention for individuals with PTSD

INTERVENTIONS:
Other: Rumination Intervention for individuals with PTSD — The intervention utilises evidence-based cognitive behavioural therapy (CBT) techniques.

SUMMARY:
After a traumatic event, it is common for thoughts to run through our minds over and over again. Typically, these include unanswerable questions like "why did this happen to me?", "what if I had done something differently?" Dwelling or ruminating on the past like this is often unhelpful and research has shown that it increases our chances of developing posttraumatic stress disorder (PTSD), a debilitating stress reaction. Once PTSD is in place, research shows that ruminating keeps the disorder going. It is unknown to what extent targeting rumination with an intervention to reduce its recurrence may help to alleviate PTSD symptoms. While rumination interventions using evidence-based cognitive behavioural therapy (CBT) have shown highly promising results in depression and anxiety research, no previous study has evaluated a stand-alone rumination intervention for individuals with PTSD.

The aim of this study is to examine the impact of a one-session online Rumination Intervention designed to reduce rumination in a small sample of 14 individuals who are currently awaiting treatment for PTSD in a British national mental health (NHS) service. The study will explore whether the Rumination Intervention reduces PTSD-related rumination, as well as PTSD and depression symptoms. It will also investigate how feasible and acceptable the intervention is for participants.

If the findings are promising, the intervention could be tested in a larger clinical study in the future. Results may help inform online interventions for PTSD.

DETAILED DESCRIPTION:
Please note: This study adopts a within and between-subjects concurrent multiple baseline A-B design will be used for this study. Due to the format of a case series, there will be no control group and no blinding. Participants will be compared to their own baseline (within) and between groups (delayed baseline for arm 2), meaning that individuals with a 3-week baseline will be compared to individuals with a 5-week baseline. This will be an experimental framework.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Willing and able to complete an online measures, online training and a phone or video call (this includes access to internet and to a computer, laptop, tablet or phone).
* Aged 18-65 years.
* English speakers and ability to read and write in English.
* Availability to participate in 6-8 weeks of this study.
* Suspected primary diagnosis of PTSD
* Currently on the waitlist for Step 3 individual PTSD treatment in an Improving Access to Psychological Therapies (IAPT) service at the Oxford Health NHS Trust or Berkshire Healthcare Foundation Trust
* Individuals must still have 9+ weeks left on the waitlist so start of PTSD treatment will not interfere with the study.
* Score above cut-off for PTSD symptoms at screening (by scoring 33 or above on the PCL-5 scores)
* Showing high rumination (by scoring "often" or "always" on any item of the RIQ)

Exclusion Criteria:

* If it appears that a different disorder/mental health condition (not PTSD) is primary (e.g. depression, substance use).
* Any other significant disease or disorder which, in the opinion of the investigators, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Weekly change of rumination: Response to Intrusion Questionnaire (RIQ; Clohessy & Ehlers, 1999; Murray et al., 2002; Steil & Ehlers, 2000) | At screening, baseline weeks 1, 2, 3, (weeks 4 & 5 for participants in 5-week baseline arm), and weeks 1 & 2 post intervention
  The RIQ is a 19-item self-report measure which examines responses to intrusive memories. It is divided into three subscales: suppression (6 items), rumination (6-8 items) and dissociation (5 items) which are scored on a scale from 0=never to 3=always. The scales have demonstrated adequate reliability and predictive validity in a range of studies (Beierl et al., 2019; Ehring, Ehlers, et al., 2008; Kleim et al., 2007). The internal consistency of the rumination subscale was between α=.80-.86. For the current study, only the 6-item rumination subscale will be used, in line with the measure recommended on the website of the Oxford Centre for Anxiety Disorder and Trauma (OxCADAT), who developed the measure. For the current study, the "high rumination" inclusion criteria was defined as individuals marking 2 (often) or 3 (always) on any of the 6 items.

SECONDARY OUTCOMES:
Weekly change of repetitive negative thinking: Repetitive Thinking Questionnaire (RTQ-10; Mahoney et al., 2012; McEvoy et al., 2010) | Baseline weeks 1, 2, 3, (weeks 4 & 5 for participants in 5-week baseline arm), and weeks 1 & 2 post intervention
  The RTQ-10 is a transdiagnostic measure of repetitive negative thinking, focused on a distressing event. Items are rated along a 5-point scale: Not at all true (1), Somewhat true (3), or Very true (5). It showed good internal consistency (α=.72-.93), convergent validity, and predictive utility in a student sample (McEvoy et al., 2010). For the current study the 10-item short form is used (Mahoney et al., 2012) instead of the longer 31-item (McEvoy et al., 2010). The short scale was highly correlated with the full scale (r=.95, p < .001) in Mahoney et al., 2012.
Weekly change of time spent ruminating | Baseline weeks 1, 2, 3, (weeks 4 & 5 for participants in 5-week baseline arm), and weeks 1 & 2 post intervention
  One-item question assessing time spent ruminating per week (estimated hours/minutes)
Weekly change of PTSD: PTSD Scale for DSM-5 (PCL-5; Blevins et al., 2015) | At screening, baseline weeks 1, 2, 3, (weeks 4 & 5 for participants in 5-week baseline arm), and weeks 1 & 2 post intervention
  The PCL-5 is a 20-item measure of PTSD symptoms directly corresponding to the DSM-5 PTSD criteria (American Psychiatric Association, 2013). Initial psychometric evaluation of the PCL-5 with university students exposed to trauma showed strong internal consistency (α=.94), and test- retest reliability (r=.82; Blevins et al., 2015). Symptoms are rated on a scale from 0=not at all to 4=extremely. A total score of 33 or more (out of a maximum score of 80) has been recommended as the preliminary clinical cut-off with higher scores indicting greater PTSD symptoms.
Pre-post change of depression: Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) | Baseline week 1 and post-intervention week 2 (pre-post measure)
  The PHQ-9 is a 9-item self-report questionnaire based on DSM-IV (American Psychiatric Association, 1994) criteria for depression. Scores range from 0=not at all to 3=nearly every day, with a score of 10 or more on the PHQ-9 indicating possible clinically significant depression with a sensitivity and specificity of 88% (Kroenke et al., 2001). Kroenke and team reported good internal reliability (α=.89) and test-retest reliability with a kappa of .84 after 48 hours.
Adherence measure | Week 2 post-intervention (end of study)
  One-item question on adherence (using the learned rumination techniques) post-intervention. The question on adherence is in line with the "acceptability" area of focus within a feasibility assessment, as recommended by Bowen and colleagues (2009).
Feasibility and acceptability measure | Week 2 post-intervention (end of study)
  Questions on feasibility and acceptability based on examples by other authors (March et al., 2018; Miner et al., 2016). Questions are in line with guidance by Bowen and colleagues on how to design feasibility studies (Bowen et al., 2009) and relate to the feasibility areas of focus of "Acceptability" and "Practicality".

OTHER OUTCOMES:
Demographic questions | At screening / pre
  Demographic questions relating to age, gender, ethnicity, time spent on waitlist, previous mental health diagnoses, and previous PTSD treatment. Ethnicity will be collected in line with guidance by the National Institute for Health and Care Research (NIHR, 2020) to include underserved and minority groups in research. By collecting data on ethnicity, research can later reflect on whether underserved and minority groups were included and, if applicable, highlight limitations of the research.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wild, BS MEd DClin, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Talking Therapies, Berkshire Healthcare NHS Foundation Trust, Bracknell, Berkshire
  - Healthy Minds, Oxford Health NHS Foundation Trust, High Wycombe